CLINICAL TRIAL: NCT03028480
Title: Nucala® Subcutaneous Injection Special Drug Use Investigation (Long-Term)
Brief Title: Long Term Special Drug Use Investigation of Mepolizumab
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 204524
Record Dates: First submitted 2017-01-06; First posted 2017-01-23 (Estimated); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Asthma
Keywords: Exacerbation; Mepolizumab; NUCALA
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with Bronchial asthma: Subjects with a refractory asthma whose symptoms are inadequately controlled despite receiving standard asthma medications will be enrolled
  Interventions: Drug: NUCALA Injection

INTERVENTIONS:
Drug: NUCALA Injection — Single dose of NUCALA SC will be administered. Dose unit, daily dose frequency, date of administration will be at the investigator discretion.

SUMMARY:
This study is a special drug use investigation program of NUCALA (a brand name for Mepolizumab) administered subcutaneously (SC). In this study the information regarding the safety and effectiveness of long term use of NUCALA after subcutaneous injection will be collected from Asthma subjects in daily clinical practice. The observation period per subject will be 52 weeks from the initiation of NUCALA treatment with follow-up investigation for 2 years after the observation period. NUCALA is a registered trademark of the GlaxoSmithKline [GSK] group of companies

ELIGIBILITY:
Inclusion Criteria:

* Subjects receiving NUCALA for the first time for treatment of bronchial asthma (a refractory asthma whose symptoms are inadequately controlled despite receiving standard asthma medications)

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects receiving NUCALA for the first time for treatment of bronchial asthma (a refractory asthma whose symptoms are inadequately controlled despite receiving standard asthma medications)
Sampling Method: Probability Sample
Enrollment: 1061 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study aims to collect and assess information regarding the safety and effectiveness of long-term use of NUCALA in asthma participants in daily clinical practice.
Pre-assignment Details: A total of 1061 participants were enrolled in the study (Enrolled Set included participants registered within the enrollment period specified in the protocol).
Groups:
- Participants With Bronchial Asthma: Participants receiving NUCALA for the first time for treatment of bronchial asthma (a refractory asthma whose symptoms were inadequately controlled despite receiving standard asthma medications) in clinical practice were enrolled in this study. No study treatment was administered during conduct of this study.
Period: Overall Study
Arm/Group | Participants With Bronchial Asthma
Started (Enrolled Set) | 1061
Safety Population | 1027
Completed | 1027
Not Completed | 34
Not completed — No revisit after the first prescription date | 2
Not completed — Did not use the drug | 1
Not completed — Violation of the enrollment deadline | 10
Not completed — Case report forms were not collected | 21

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for the Safety Analysis Set which consisted of the participants fixed in the case report form. It includes participants that do not fall under the safety analysis exclusion criteria.
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 1027
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 641
  Male | 386
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1027
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Data Entered on Electronic Data Capture (EDC) System
Description: The number of participants whose data was entered in the EDC system up to 14 days from the initiation of NUCALA treatment (Day 1) has been presented.
Time Frame: Up to 14 days from the initiation of NUCALA treatment (Day 1)
Population: Enrolled Set included participants registered within the enrollment period specified in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 1061
Participants | 1040

2. Primary Outcome: Percentage of Participants With Adverse Drug Reaction (ADR)
Description: ADR is defined as a response to a drug which is noxious and unintended, and which occurred at doses normally used in man for the prophylaxis, diagnosis, or therapy of disease, or for the modifications of physiological function. Percentage of participants with ADR were calculated as the number of participants having a particular ADR divided by total number of participants on NUCALA treatment*100. Percentage values are rounded-off.
Time Frame: Up to 3 years
Population: Safety Analysis Set consisted of the participants fixed in the case report form (CRF). It included participants that do not fall under the safety analysis exclusion criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 1027
Percentage of participants | 4.1

3. Primary Outcome: Number of Participants Showing Response to the Treatment
Description: The number of participants who showed response to the bronchial asthma treatment has been presented.
Time Frame: Up to 1 year
Population: Effectiveness Analysis Set consisted of the participants included in safety analysis, participants that do not fall under the participants excluded from efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 959
Participants | 866

4. Primary Outcome: Number of Participants Excluded From Analysis Due to Exacerbation of Asthma
Description: The number of participants excluded from analysis due to exacerbation of asthma has been presented.
Time Frame: Up to 1 year
Population: Enrolled Set included participants registered within the enrollment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 1061
Participants | 16

5. Primary Outcome: Number of Participants With Adverse Drug Reactions (ADR)
Description: ADR is defined as a response to a drug which is noxious and unintended, and which occurred at doses normally used in man for the prophylaxis, diagnosis, or therapy of disease, or for the modifications of physiological function.
Time Frame: Up to 3 years
Population: Safety Analysis Set consisted of the participants fixed in the case report form. It included participants that do not fall under the safety analysis exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 1027
Participants | 42

6. Primary Outcome: Percentage of Participants With Occurrences of Safety Specifications and Priority Investigation Matters
Description: Safety specifications and priority investigation matters included hypersensitivity reaction including anaphylaxis, infections, and malignant tumor. The percentage of participants with occurrences of safety specifications and priority investigation matters have been reported. Percentage values are rounded-off.
Time Frame: Up to 3 years
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 1027
Percentage of participants
  Hypersensitivity reaction including anaphylaxis | 1.2
  Infections | 0.3
  Malignant tumor | 0.2

7. Secondary Outcome: Response Rate Assessed by Global Assessment of Effectiveness
Description: Response rate is the percentage of participants assessed as "effective" based on the course of subjective symptoms and clinical symptoms. Response rate was calculated as number of participants showing response to the NUCALA treatment divided by total number of participants on treatment*100. Percentage values are rounded-off. Response rate and corresponding 95% confidence interval were reported.
Time Frame: Up to 1 year
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 959
Percentage of participants | 90.3 [88.3 to 92.1]

8. Secondary Outcome: Rate of Exacerbation of Asthma
Description: Asthma exacerbation was defined as new or increased asthma symptoms (wheezing, coughing, dyspnea, chest tightness, and/or nighttime awakenings due to these symptoms) that resulted in hospitalization, emergency room visit and usage of systemic steroids. Exacerbation rate was defined as number of asthma exacerbations divided by total person-year (52 weeks were converted to 1 year). Data for exacerbations requiring hospitalization, emergency room visit, and use of systemic corticosteroid have been presented.
Time Frame: 52 weeks before the initiation of NUCALA treatment (Day 1) and at Week 52 post-treatment
Population: Effectiveness Analysis Set consisted of the participants included in safety analysis, participants that do not fall under the participants excluded from efficacy analysis. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Number; unit: Asthma exacerbations per person-year
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 959
Asthma exacerbations per person-year
  Exacerbations requiring hospitalization: 52 weeks before the initiation of NUCALA treatment: number analyzed (Participants) | 956
  Exacerbations requiring hospitalization: 52 weeks before the initiation of NUCALA treatment | 0.4
  Exacerbations requiring hospitalization: at Week 52 post-treatment | 0.1
  Exacerbations requiring emergency room visits: 52 weeks before the initiation of NUCALA treatment: number analyzed (Participants) | 943
  Exacerbations requiring emergency room visits: 52 weeks before the initiation of NUCALA treatment | 0.9
  Exacerbations requiring emergency room visits: at Week 52 post-treatment | 0.2
  Exacerbations requiring use of systemic corticosteroid:52weeks before initiation of NUCALA treatment: number analyzed (Participants) | 956
  Exacerbations requiring use of systemic corticosteroid:52weeks before initiation of NUCALA treatment | 3.2
  Exacerbations requiring the use of systemic corticosteroid: at Week 52 post-treatment | 0.7

9. Secondary Outcome: Total Score of Asthma Control Test (ACT) at Indicated Time Points
Description: The ACT is a validated self-completed questionnaire utilizing 5 questions to assess asthma control on a 5-point categorical scale ranging from 1 (not controlled at all) to 5 (completely controlled) with higher scores indicating better control. Total ACT score is calculated as the sum of the scores from the 5 questions and can range from 5 to 25, with higher scores indicating better control. An ACT total score of 5 to 19 suggests that the participant's asthma is unlikely to be well controlled, whilst a score of 20 to 25 suggests that the participant's asthma is likely to be well controlled. Baseline was defined as within 8 weeks prior to initiation of NUCALA treatment (Day 1).
Time Frame: Baseline, Weeks 12, 24 and 52 after the initiation of NUCALA treatment (Day 1)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 352
Scores on a scale
  Baseline | 16.2 (4.9)
  12 weeks after the initiation of NUCALA treatment: number analyzed (Participants) | 317
  12 weeks after the initiation of NUCALA treatment | 20.5 (4.3)
  24 weeks after the initiation of NUCALA treatment: number analyzed (Participants) | 261
  24 weeks after the initiation of NUCALA treatment | 20.9 (4.2)
  52 weeks after the initiation of NUCALA treatment: number analyzed (Participants) | 221
  52 weeks after the initiation of NUCALA treatment | 21.4 (4.0)

10. Secondary Outcome: Mean Peak Expiratory Flow (PEF) at Indicated Time Points
Description: Peak Expiratory Flow is a person's maximum speed of expiration. PEF was measured using an electronic peak expiratory flow device (ePEF) at Baseline (Day 1), and at Weeks 12, 24, and 54 after the initiation of NUCALA treatment. Baseline was defined as within 8 weeks prior to initiation of NUCALA treatment (Day 1).
Time Frame: Baseline, Weeks 12, 24 and 52 after the initiation of NUCALA treatment (Day 1)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Participants With Bronchial Asthma
Number analyzed (Participants) | 120
Liters/minute
  Baseline | 304.4 (146.8)
  12 weeks after the initiation of NUCALA treatment: number analyzed (Participants) | 78
  12 weeks after the initiation of NUCALA treatment | 333.7 (150.5)
  24 weeks after the initiation of NUCALA treatment: number analyzed (Participants) | 51
  24 weeks after the initiation of NUCALA treatment | 334.2 (138.7)
  52 weeks after the initiation of NUCALA treatment: number analyzed (Participants) | 45
  52 weeks after the initiation of NUCALA treatment | 358.9 (129.8)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and non-serious adverse drug reactions (ADRs) were collected up to 3 years
Description: All-cause mortality, serious and non-serious ADRs were reported for Safety Analysis Set (1027) since 34 participants from Enrolled Set (1061) were not included in safety analysis as their CRF were not collected/fall under safety analysis exclusion criteria. Safety Analysis Set consisted of participants fixed in CRF. It includes participants that do not fall under safety analysis exclusion criteria. Only serious and non-serious ADR were collected but not all adverse events as planned per Protocol
Arm/Group | Participants With Bronchial Asthma
All-Cause Mortality (participants affected / at risk) | 3/1027
Serious Adverse Events (participants affected / at risk) | 9/1027
Other Adverse Events (participants affected / at risk) | 33/1027
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Bronchial Asthma (N=1027)
Pneumonia (Infections and infestations) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myasthenia gravis (Nervous system disorders) | 1
Optic neuropathy (Eye disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Chronic eosinophilic rhinosinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Condition aggravated (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Bronchial Asthma (N=1027)
Bronchitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Headache (Nervous system disorders) | 2
Palpitations (Cardiac disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Chronic eosinophilic rhinosinusitis (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Condition aggravated (General disorders) | 3
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Eosinophil count increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT03028480/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT03028480/SAP_001.pdf